### **Masonic Cancer Center, University of Minnesota**

#### SCREENING CONSENT

Phase I/II Study of Human Chorionic Gonadotropin and Epidermal Growth Factor Supplementation (Pregnyl®) to Support Tolerance and Repair As Adjunct Therapy in High-Risk or Refractory Acute Graft-Versus-Host Disease

High-risk aGVHD - ARM 1

Principal Investigator:
Shernan G. Holtan, MD
Division of Hematology, Oncology and Transplantation

For questions about research appointments, the research study, research results, or other concerns, contact the study team at:

Lead Investigator: Dr. Shernan Holtan

Phone Number: (612) 301-1095 Email Address: sgholtan@umn.edu

The study will be conducted at 2 cancer research centers around the United States; however the University of Minnesota is the lead institution and Shernan Holtan, MD from Hematology, Oncology and Transplantation is the principal investigator (the physician in charge) of this research study. Up to 88 patients will be treated on this study nationally: 78 at the University of Minnesota and 10 at Rush University in Chicago, IL.

You are invited to participate in this research study because you have acute Graft-Versus-Host Disease (GVHD), a complication of your recent hematopoietic cell transplant. To be considered for this study you must be between the ages of 0 and 76 years and have acute GVHD which, because of its severity, is at a high-risk of not being controlled by the usual therapy alone.

You may be eligible for a therapy for GVHD that involves using a drug called Pregnyl, also known as hormone human chorionic gonadotropin (HCG). Pregnyl is approved by

January 29, 2020


Affix Donor Label Here

MT2014-12: Screening Consent - ARM 1

the United States Food and Drug Administration (FDA) to treat infertility in women by stimulating ovulation as well as to treat testicle development issues in males. Its use in acute GVHD is considered investigational.

However, before doing a full evaluation, we are requesting permission to do some pretesting on a blood sample to see if you have a specific biomarker in your blood. A biomarker is a measureable substance in your body that is a sign or a predictor of whether or not you have a disease, or how a disease may react to therapy. The biomarker we are looking for in this case, amphiregulin, is a protein that can be used to define your risk for GVHD.

You are asked to read this form before you agree to the pre-screening process. If you have any questions, we will make sure they are answered before you agree.

If you agree by signing this consent form, a blood sample will be collected.

The pre-screening blood sample will be tested as follows:

Your blood will be tested for the **amphiregulin biomarker**.

The biomarker will help determine whether or not you may be eligible for this study and/or which part of the study treatment may be the most beneficial.

**Risks** 

You will have slightly less than 1 tablespoon of blood collected. The risks of having **blood drawn** include pain, bruising and/or redness where the blood is drawn from your arm. Rarely this place where the needle is stuck in becomes infected (red, warm, swelling). Some people feel faint (like they may pass out) when having blood drawn, but this can be avoided by looking away.

**Benefits** 

There will be no benefit to you for the pre-screening. You will not be paid.

Costs

The costs of this lab test is paid for by the study.

January 29, 2020


## **Research Related Injury**

In the event that this research activity results in an injury, treatment is available, including first aid, emergency treatment and follow-up care as needed. Care for such injuries will be billed in the ordinary manner to you or your insurance company. If you think you have suffered a research related injury, let someone associated with the study know right away.

## Confidentiality

The records of this study will be kept private. Information gained from this study will be used for research and educational purposes. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used.

Organizations that may look at and/or copy your medical record for research, quality assurance, and data analysis include:

- Departments at the University of Minnesota with appropriate regulatory oversight
- The National Cancer Institute (NCI) and other government agencies, like the Food and Drug Administration (FDA), involved in keeping research safe for people To this extent, confidentiality is not absolute.

A description of this clinical trial will be available at http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

#### **Use Of Identifiable Health Information**

Your PHI created or received for the purposes of this study is protected under the federal regulation known as HIPAA. Refer to the attached HIPAA authorization for details concerning the use of this information.

# **Right To Say No**

The decision to have your blood pre-screened is completely up to you. If you do not want to be considered for this study, you have the right to say no.

January 29, 2020 

MT2014-12: Screening Consent - ARM 1

#### **Contacts and Questions**

Information for contacting the study Principal Investigator is provided on the 1<sup>st</sup> page of this document.

This research has been reviewed and approved by an Institutional Review Board (IRB) within the Human Research Protections Program (HRPP). To share feedback privately with the HRPP about your research experience, call the Research Participants' Advocate Line at 612-625-1650 or go to www.irb.umn.edu/report.html. You are encouraged to contact the HRPP if:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You want to talk to someone besides the research team.
- You have questions about your rights as a research participant.
- You want to get information or provide input about this research.

#### **FEEDBACK**

After the study, you may be asked to complete a survey about your experience as a research participant. You do not have to complete the survey if you do not want to. If you do choose to complete the survey, your responses will be anonymous.

If you are not asked to complete a survey after the study is over, but you would like to share feedback, please contact the study team or the Human Research Protection Program (HRPP). See the "Contacts and Questions" section of this form for study team and HRPP contact information.

January 29, 2020


Affix Donor Label Here

| ent – ARM 1 | |
|---|---|
| <b>nt</b><br>en read to me. I have had my q<br>tested as a pre-screening for a | • |
| lly authorized representative | Date |
| egally authorized representative | Э |
| er obtaining consent | Date |
| archer obtaining consent | |
| ole to read or sign this consen | t form because of the following |
| le to read the information<br>ally impaired<br>English speaking<br>ically unable to sign the consen | t form. Please describe: |
| | en read to me. I have had my contested as a pre-screening for a lily authorized representative egally authorized representative er obtaining consent er obtaining consent ele to read or sign this consent ele to read the information ally impaired english speaking ically unable to sign the consent english english speaking ically unable to sign the consent english |

Affix Donor Label Here

| MT2014-12: Screening Consent – ARM 1 | |
|---|---|
| For the Consent of Non-English Speaking Participals As someone who understands both English and the represent that the English version of the consent form in the subject's own language, and that the subject questions. | e language spoken by the subject, I<br>n was presented orally to the subject |
| Signature of Interpreter | <br>Date |
| Printed Name of Interpreter | _ |
| OR: | |
| Statement from a Non-Interpreter: As someone who understands both English and the represent that the English version of the consent form in the subject's own language, and that the subject questions. | m was presented orally to the subject |
| Signature of Individual | <br>Date |
| Printed Name of Individual | |

January 29, 2020

